CLINICAL TRIAL: NCT03218969
Title: Treatment of Restless Leg Syndrome (RLS) Augmentation With Ecopipam, a D1 Specific Antagonist
Acronym: RLS-Ecopipam
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: William Ondo, MD (Other)
Collaborators: Restless Legs Syndrome Foundation (Unknown)
Responsible Party: Sponsor-Investigator, William Ondo, MD, HMRI Principal & Sponsor Investigator: Ondo, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro#00016705
Record Dates: First submitted 2017-04-21; First posted 2017-07-17 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Restless Legs Syndrome; Augmentation
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ecopipam

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study period 1 (Experimental): * Ecopipam or matching placebo 25 mg by mouth for 7 days (week 1), followed by
  * Ecopipam or matching placebo 50 mg by mouth for 7 days (week 2), followed by
  * Ecopipam or matching placebo 100 mg by mouth for 23 days (weeks 3).
  Interventions: Drug: Ecopipam; Drug: Placebo
- Study period 2 (Experimental): * Matching placebo or ecopipam 25 mg by mouth for 7 days (week 7), followed by
  * Matching placebo or ecopipam 50 mg by mouth for 7 days (week 8), followed by
  * Matching placebo or ecopipam 100 mg by mouth for 23 days (week 9).
  Interventions: Drug: Ecopipam; Drug: Placebo

INTERVENTIONS:
Drug: Ecopipam — oral drug in subjection currently experiencing dopamine agonist induced augmentation
  Other Names: PSYRX101
Drug: Placebo — matching placebo

SUMMARY:
This is an exploratory, double blinded cross-over study of the D1 antagonist ecopipam treat patients currently having dopamine agonist induced augmentation in restless legs syndrome. Each arm is 6 weeks composed of an unforced titration up to 100mg/day separated by a 2-week wash-out period. Efficacy points will include the IRLS, augmentation scales, sleep scales, clinical impressions and fatigue/mood scales.

DETAILED DESCRIPTION:
This is a double-blind, exploratory proof of concept, cross-over trial of the D1 antagonist ecopipam for subjects with augmented Restless legs syndrome (RLS). Investigators will recruit 10 subjects taking dopamine agonists for RLS who are currently experiencing augmentation. The goal is to have 8 completers. There is no power analysis as this is an exploratory study and there is no previous data on treatment of augmentation. "Meaningful improvement" is not even established. A safety analysis will be done after 5 subjects have been enrolled. Duration of study and is based mostly on contracted drug availability for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Provide consent to participate in the study
* Individuals of either sex, 21-80 years of age
* Clinically defined Restless Leg Syndrome, and problematic augmentation currently on monotherapy with dopaminergic treatment.

Exclusion Criteria:

* Current use of Opioid medications
* Clinical relevant depression or other medical problems that in the opinion of the investigator would not allow for safe completion of the protocol.
* Suicidal ideation
* History of epilepsy
* Current MAO inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-10-15 (Estimated)

PRIMARY OUTCOMES:
International RLS Rating scale | baseline to end of each treatment arm (6 weeks)
  scale
Augmentation severity scale | baseline to end of each treatment arm (6 weeks)
  scale

SECONDARY OUTCOMES:
24 hour RLS diary | Day 0 (visit 1) to end of each treatment arm (6 weeks)
  diary of RLS symptoms
Clinical Global Impression | From start of each treatment arm through one week after treatment withdrawal
  scale

OTHER OUTCOMES:
Hamilton depresion scale | baseline to end of each treatment arm (6 weeks)
  scale
MOS sleep scale | baseline to end of each treatment arm (6 weeks)
  scale
Fatigue severity scale | baseline to end of each treatment arm (6 weeks)
  scale
Columbia Suicide Severity Rating Scale | baseline to end of each treatment arm (6 weeks)
  scale
Epworth sleep scale | baseline to end of each treatment arm (6 weeks)
  scale
Serum chemistry (liver enzymes ALT and AST) | baseline to end of each treatment arm (6 weeks)
  safety assessment
Vital signs | baseline to end of each treatment arm (6 weeks)
  safety assessment
Physical/Neurological exam | baseline to end of each treatment arm (6 weeks)
  safety assessment
12 lead ECG | baseline to end of each treatment arm (6 weeks)
  safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: William G. Ondo, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided